CLINICAL TRIAL: NCT03471299
Title: Impact of Ultrafiltration Rates on Mortality in Maintenance Hemodialysis Patients
Brief Title: Association of Survival in Impact of Ultrafiltration Rates in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: University of Hyogo (Other)
Responsible Party: Principal Investigator, Yoshihiro Tsuji, clinical engineer, University of Hyogo
Other Study IDs: Uhyogo3
Record Dates: First submitted 2018-03-13; First posted 2018-03-20 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Hemodialysis
Keywords: Ultrafiltration rate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study assesses retrospectively the association of mortality on UFR assessments in our study population undergoing HD.

ELIGIBILITY:
Inclusion Criteria:

Patients with stable undergoing hemodialysis for >1 year.

Exclusion Criteria:

Patients with combined therapy with peritoneal dialysis and HD. Patients without records of laboratory investigations during this period. Patients with transferred hospital and those lost to follow-up.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: In this study, 759 patients who had undergone maintenance HD for >1 year at Tojinkai Hospital, kyoto, Japan. The present study examined data from all individual with regular thrice weekly maintenance HD treatment.
Sampling Method: Probability Sample
Enrollment: 759 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Ultrafiltration rate (ml/hr/kg) | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Yuko Mizuno-Matsumoto, Ph.D, Study Director — Graduate School of Applied Informatics, University of Hyogo
Locations (1):
- Graduate School of Applied Informatics, University of Hyogo, Kobe, Hyōgo, Japan